CLINICAL TRIAL: NCT00807456
Title: A Prospective, Open, Single Arm, Multi-center Study to Evaluate Maintenance of Lingual Bone in Healed Ridges With the ASTRA TECH Implant System, OsseoSpeed™ Profile Implant. A 3-year Follow-up Study
Brief Title: Study to Evaluate an Implant With a Sloped Top in Patients With a Sloped Jaw Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-PRO-0001
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects treated with ASTRA TECH Implant System, OsseoSpeed™ Profile implant (Experimental)
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™

INTERVENTIONS:
Device: ASTRA TECH Implant System, OsseoSpeed™ — ASTRA TECH Implant System, OsseoSpeed™ Profile implants: Ø4.5, 5.0, 5.0S mm in lengths of 9, 11, 13, 15mm.

SUMMARY:
The study aims to evaluate maintenance of lingual/palatinal marginal bone with the (ASTRA TECH Implant System) OsseoSpeed™ Profile implant in sites where the alveolar crest anatomy is sloped in a lingual to buccal direction.

The hypothesis is that the sloped marginal contour of the implant will help preserve the lingual/palatinal marginal bone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Aged 18-75 years at enrolment
* A lingual-buccal difference in bone height between 2.0-5.0 mm at the implant site
* History of edentulism in the study area of at least 3 months
* Presence of alveolar bone crest dimensions judged by the investigator to allow ≥1mm of bone circumferential to the implant after implant placement.
* In need for a single implant replacing a missing tooth in any location with an adjacent natural tooth mesially, and an adjacent natural tooth or edentulous space distally to the planned implant position (i.e. no existing or planned implant adjacent to the planned study implant position)
* Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

* Uncontrolled pathological processes in the oral cavity
* Known or suspected current malignancy
* History of radiation therapy in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Uncontrolled diabetes mellitus
* Corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Smoking more than 10 cigarettes per day
* Present alcohol and/or drug abuse
* Current need for bone grafting in the planned implant area
* Previous enrolment in the present study
* Simultaneous participation in another clinical study or participation in a clinical study during the last 6 months
* Involvement in the planning and conduct of the study (applies to both Sponsor staff or staff at the study site)
* Unlikely to be able to comply with study procedures, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, Prof., Study Chair — Department of Periodontology, Sahlgrenska Academy at University of Gothenburg
Locations (5):
- United States (2):
  - Department of Periodontology, College of Dental Medicine, Nova Southeastern University, Fort Lauderdale, Florida
  - Department of Periodontics, Robert Schattner Center, School of Dental Medicine, University of Pennsylvania, Philadelphia, Pennsylvania
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - Praxis Dr Robert Nölken, Lindau
- Studio Dentistico Donati, Perugia, Italy

REFERENCES:
- [Result] Noelken R, Donati M, Fiorellini J, Gellrich NC, Parker W, Wada K, Berglundh T. Soft and hard tissue alterations around implants placed in an alveolar ridge with a sloped configuration. Clin Oral Implants Res. 2014 Jan;25(1):3-9. doi: 10.1111/clr.12079. Epub 2012 Dec 5. PMID 23210667

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Treated With OsseoSpeed™ Profile Implant: ASTRA TECH Implant System, OsseoSpeed™: ASTRA TECH Implant System, OsseoSpeed™ Profile implants: Ø4.5, 5.0, 5.0S mm in lengths of 9, 11, 13, 15mm.
Period: Overall Study
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Started | 65
Surgical Re-entry (Implant Placement + 16-17 Weeks) | 65
Completed | 57
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Treated With ASTRA TECH Implant System, OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.05 (13.974)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Bone Level Changes at the Lingual Aspect From Implant Placement (Baseline) to Re-entry 16 Weeks After Implant Placement
Description: Clinical measurements after implant installation and after 16 weeks to determine bone levels at the buccal and lingual aspects in relation to a fixed landmark on the implant, i.e. the interface between the micro-threaded part and the shoulder at the marginal portion of the implants.The assessments were made using a periodontal probe and distances were measured to the nearest 0.5 mm. Negative value denotes loss of bone.
Time Frame: At baseline and 16 weeks
Population: Per-protocol analysis set
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 65
Number analyzed (Implants) | 65
mm | -0.02 (0.49)

2. Secondary Outcome: Implant Survival Rate
Description: The survival rate for individual implants was evaluated at each visit. Any removed implant was considered an implant loss, regardless of reason for removal.
Time Frame: 21 weeks, 12 months, 24 months and 36 months post implant placement.
Population: Per-protocol analysis set
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Groups:
- Subjects Assessed at Permanent Restoration 21 Weeks Post Implant Placement; Subjects Assessed at 12 Months Post Implant Placement; Subjects Assessed at 24 Months Post Implant Placement; Subjects Assessed at 36 Months Post Implant Placement: Subjects treated with ASTRA TECH Implant System, OsseoSpeed™: ASTRA TECH Implant System, OsseoSpeed™ Profile implants: Ø4.5, 5.0, 5.0S mm in lengths of 9, 11, 13, 15mm.
Arm/Group | Subjects Assessed at Permanent Restoration 21 Weeks Post Implant Placement | Subjects Assessed at 12 Months Post Implant Placement | Subjects Assessed at 24 Months Post Implant Placement | Subjects Assessed at 36 Months Post Implant Placement
Number analyzed (Participants) | 65 | 64 | 59 | 57
Number analyzed (Implants) | 65 | 64 | 59 | 57
Implants | 65 | 64 | 59 | 57

3. Secondary Outcome: Marginal Bone Level (MBL) Change From Implant Placement Presented on Implant Level
Description: MBL alteration assessed by measuring the distance from the implant reference point to the most conical bone-to-implant contact on the mesial and distal side of the implant. The mean of all values for one subject was calculated and used for analysis.
Time Frame: Baseline and 16 weeks, 21 weeks, 12 months, and 36 months post implant placement
Population: Per-protocol analysis set. All subjects/implants available for each visit are included in below analyses.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 56
Number analyzed (Implants) | 56
mm
  Implant Placement to re-entry (implant placement + 16 weeks) | -0.28 (0.68)
  Implant placement to permanent restoration (implant placement + 21 weeks): number analyzed (Participants) | 55
  Implant placement to permanent restoration (implant placement + 21 weeks): number analyzed (Implants) | 55
  Implant placement to permanent restoration (implant placement + 21 weeks) | -0.48 (0.74)
  Implant placement to implant placement + 12 months: number analyzed (Participants) | 55
  Implant placement to implant placement + 12 months: number analyzed (Implants) | 55
  Implant placement to implant placement + 12 months | -0.29 (1.10)
  Implant placement to implant placement + 36 months: number analyzed (Participants) | 52
  Implant placement to implant placement + 36 months: number analyzed (Implants) | 52
  Implant placement to implant placement + 36 months | -0.57 (1.60)

4. Secondary Outcome: Condition of Peri-Implant Tissues Measured Through Bleeding on Probing (BoP)
Description: BoP was assessed by recording bleeding after probing at the mesial, distal, buccal, and palatal surfaces of the implant site.
Time Frame: 21 weeks, 12 months, 24 months, and 36 months post implant placement
Population: Per-protocol analysis set. All subjects available for each visit are included in below analyses.
Measure: Number; unit: Implants with BoP
Units Other Than Participants: Implants
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 65
Number analyzed (Implants) | 65
Implants with BoP
  Permanent restoration 21 weeks after implant placement | 2
  12 months after implant placement: number analyzed (Participants) | 64
  12 months after implant placement: number analyzed (Implants) | 64
  12 months after implant placement | 20
  24 months after implant placement: number analyzed (Participants) | 59
  24 months after implant placement: number analyzed (Implants) | 59
  24 months after implant placement | 16
  36 months after implant placement: number analyzed (Participants) | 57
  36 months after implant placement: number analyzed (Implants) | 57
  36 months after implant placement | 21

5. Secondary Outcome: Condition of Peri-implant Tissues Measured by Average Change in Probing Pocket Depth (PPD) From Permanent Restoration
Description: PPD was measured using a regular peridontal probe from the gingival margin to nearest whole millimeter. The average PPD change from permanent restoration is presented on implant level.
Time Frame: Baseline and 12 months, 24 months, and 36 months post implant placement
Population: Per-protocol analysis set. All subjects available for each visit are included in below analyses.
Measure: Mean (Standard Deviation); unit: PPD in mm
Units Other Than Participants: Implants
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 63
Number analyzed (Implants) | 63
PPD in mm
  Permanent restoration to 12 months post implant placement | 0.28 (0.73)
  Permanent restoration to 24 months post implant placement: number analyzed (Participants) | 58
  Permanent restoration to 24 months post implant placement: number analyzed (Implants) | 58
  Permanent restoration to 24 months post implant placement | 0.31 (0.68)
  Permanent restoration to 36 months post implant placement: number analyzed (Participants) | 57
  Permanent restoration to 36 months post implant placement: number analyzed (Implants) | 57
  Permanent restoration to 36 months post implant placement | 0.36 (0.85)

6. Secondary Outcome: Condition of Peri-implant Tissues Measured by Average Change in Clinical Attachment Level (CAL) From Permanent Restoration
Description: CAL was measure with a probe from the crown margin (the interface between the abutment) to the crown at the mesial, buccal, distal, and lingual aspects of the implant. The average CAL change from permanent restoration is presented on implant level.
Time Frame: Baseline and 12 months, 24 months, and 36 months post implant placement
Population: Per-protocol analysis set. All subjects available for each visit are included in below analyses.
Measure: Mean (Standard Deviation); unit: CAL in mm
Units Other Than Participants: Implants
Arm/Group | Subjects Treated With OsseoSpeed™ Profile Implant
Number analyzed (Participants) | 63
Number analyzed (Implants) | 63
CAL in mm
  Permanent restoration to 12 months post implant placement | 0.02 (0.54)
  Permanent restoration to 24 months post implant placement: number analyzed (Participants) | 58
  Permanent restoration to 24 months post implant placement: number analyzed (Implants) | 58
  Permanent restoration to 24 months post implant placement | 0.14 (0.57)
  Permanent restoration to 36 months post implant placement: number analyzed (Participants) | 57
  Permanent restoration to 36 months post implant placement: number analyzed (Implants) | 57
  Permanent restoration to 36 months post implant placement | 0.11 (0.85)

ADVERSE EVENTS:
Time Frame: Up to 3 years post implant placement
Groups:
- ASTRA TECH Implant System, OsseoSpeed™ Profile: ASTRA TECH Implant System, OsseoSpeed™: ASTRA TECH Implant System, OsseoSpeed™ Profile implants: Ø4.5, 5.0, 5.0S mm in lengths of 9, 11, 13, 15mm.
Arm/Group | ASTRA TECH Implant System, OsseoSpeed™ Profile
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 2/65
Other Adverse Events (participants affected / at risk) | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASTRA TECH Implant System, OsseoSpeed™ Profile (N=65)
Hip surgery (Surgical and medical procedures) | 1 (1)
Melanoma (Skin and subcutaneous tissue disorders) | 1 (1) — Skin cancer left ring finger

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less